CLINICAL TRIAL: NCT04827745
Title: A Multicenter Phase II Study of Blinatumomab for Treatment of Adult Patients With Morphologic Relapsed/Refractory or Measurable Residual Disease (MRD) CD19-Positive Mixed Phenotype Acute Leukemia (MPAL)
Brief Title: Blinatumomab for Treatment of R/R or MRD-positive CD19-Positive MPAL
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2099GCCC ; HP-00094794
Record Dates: First submitted 2021-03-25; First posted 2021-04-01 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-07

CONDITIONS: Mixed Phenotype Acute Leukemia (MPAL); Measurable Residual Disease (MRD)
MeSH Terms: conditions — Leukemia, Biphenotypic, Acute; Neoplasm, Residual | interventions — blinatumomab

STUDY DESIGN:
Intervention Model Description: Cohort A: Subjects with R/R CD19-positive MPAL
  CohortB: Subjects with CD19-positive MPAL in complete remission and detectable MRD
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Subjects with R/R CD19-positive MPAL (Experimental): Cohort A: Evaluate the efficacy of blinatumomab to achieve the best morphologic response after the first two cycles of therapy in subjects with morphologic R/R CD19-positive MPAL
  * The treatment of blinatumomab consists of induction, consolidation and maintenance therapy
  * Subject will receive study drug blinatumomab by continuous IV infusion (CIV)
  * Each treatment cycle consists of 28 days of blinatumomab CIV followed by a 14±3 days treatment-free interval for induction, 28±3 days treatment-free interval for consolidation, and 56±3 days treatment-free interval for maintenance
  * The initial dose of blinatumomab is 9 mcg/day for 7 days. The target dose for rest of treatment is 28 mcg/day
  Interventions: Drug: BLINCYTO (Blinatumomab)
- Subjects with CD19-positive MPAL in CR/CRh/CRi/CRp and detectable MRD (Experimental): Cohort B: Evaluate the efficacy of blinatumomab to achieve MRD-negativity in subjects with CD19-positive MPAL in CR, or CRh, or CRi or CRp after receiving at least one chemotherapy block of standard ALL or AML treatment with MRD-positivity at a level of ≥ 0.1% using an assay with a minimum sensitivity of 0.01%
  * The treatment of blinatumomab consists of induction, consolidation and maintenance therapy
  * Subject will receive study drug blinatumomab by continuous IV infusion (CIV)
  * Each treatment cycle consists of 28 days of blinatumomab CIV followed by a 14±3 days treatment-free interval for induction, 28±3 days treatment-free interval for consolidation, and 56±3 days treatment-free interval for maintenance.
  * The dose of blinatumomab is 28 mcg/day
  Interventions: Drug: BLINCYTO (Blinatumomab)

INTERVENTIONS:
Drug: BLINCYTO (Blinatumomab) — Blinatumomab (BLINCYTO , AMG 103, formerly also known as MT103 or bscCD19xCD3) is a novel single chain antibody construct in the class of the bispecific T-cell engager (BiTE®). Blinatumomab directs CD-3 positive effector memory T cells to CD19-positive target cells (Hoffmann et al, 2005; Dreier et al, 2002). The targeted CD19 antigen is constitutively expressed on normal B cells throughout a person's lifetime (Smet et al, 2011) and is highly conserved in B-cell malignancies (Tedder, 2009; Wang et al, 2012).

SUMMARY:
This is a research study to find out if a drug called blinatumomab is effective for treating patients with relapsed or refractory (R/R) or measurable residual disease (MRD) CD19-positive mixed phenotypic acute leukemia (MPAL). Measurable Residual Disease (MRD) means that there are a small number of cancer cells remaining after treatment

DETAILED DESCRIPTION:
This is a multicenter, non-randomized, open-label, phase II study evaluating the efficacy of blinatumomab to achieve the following objectives:

1. The best morphologic response after the first two cycles of therapy in subjects with morphologic R/R CD19-positive MPAL
2. MRD-negativity in subjects with CD19-positive MPAL in CR, or CRh, or CRi or CRp after receiving at least one chemotherapy block of standard ALL or AML treatment with MRD-positivity at a level of ≥ 0.1% using an assay with a minimum sensitivity of 0.01%

The trial consists two groups (Group A and B) and three phases ( induction, consolidation and maintenance) of therapy. Subject will receive study drug blinatumomab by continuous IV infusion (CIV). Each treatment cycle consists of 28 days of blinatumomab CIV followed by a 14±3 days treatment-free interval for induction, 28±3 days treatment-free interval for consolidation, and 56±3 days treatment-free interval for maintenance

Blinatumomab is approved by Food and Drug Administration [FDA] and European Medicines Agency [EMA] for use in people with another type of acute leukemia called acute lymphoblastic leukemia (ALL) but not MPAL.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have histologically or cytologically confirmed R/R CD19-positive MPAL based on the WHO criteria, OR CD19-positive MPAL in CR/CRh/CRi/CRp after at least one chemotherapy block of standard ALL or AML therapy with detectable MRD ≥ 0.1%. Primary refractory MPAL is defined by absence of CR/CRh/CRi/CRp after at least one cycle of standard AML/ALL induction therapy. A patient has relapsed MPAL if they achieved a CR/CRh/CRi/CRp after induction therapy (CR1) and has then relapsed during, or after continuation of therapy.
* Age 18 years and older
* Subjects who have undergone allo-HSCT are eligible if they are ≥ 4 weeks post stem cell infusion, have no evidence of GVHD > Grade 2, and are at least ≥ 1 week off all immunosuppressive therapy
* Previous cytotoxic chemotherapy (except for hydroxyurea) must have been completed at least 2 weeks prior to day 1 of treatment on the study. Subjects with hematologic malignancies are expected to have hematologic abnormalities at study entry.
* ECOG performance status < 3
* Subjects must have organ function as below:

  * Direct bilirubin ≤ 2.5 mg/dL
  * AST/ALT/Alkaline phosphatase ≤ 5 X institutional upper limit of normal
  * Serum creatinine ≤ 3 mg/dL
* Subjects with a history of CNS leukemia must be clinically stable with a flow cytometric clear CSF in the 2 weeks prior to day 1 of blinatumomab administration. Subjects with history of CNS leukemia in Cohort A should have received one dose of intrathecal chemotherapy in the 4 weeks prior to day 1 of blinatumomab administration. Subject can receive subsequent prophylactic intrathecal chemotherapy.
* Female subjects of childbearing potential must have a negative pregnancy test
* Ability to understand and willingness to sign a written informed consent document
* Agree to comply with the study requirements and agree to come to the clinic/hospital for required study visits

Exclusion Criteria:

* Subjects receiving any other investigational agents, or concurrent chemotherapy, radiation therapy, or immunotherapy not including corticosteroids or hydroxyurea
* Subjects with acute leukemia with any of the following cytogenetic abnormalities:

  t(15;17)(q24;q21) PML/RARA, t(8;21)(q22;q22) RUNX1/RUNX1T1, inv(16)(p13q22)/t(16;16)(p13;q22) CBFB-MYH11
* A history or presence of clinically relevant CNS pathology (e.g., as epilepsy, paresis, aphasia, stroke, severe brain injuries, dementia, cerebellar disease, psychosis)
* Hyperleukocytosis with > 50,000 blasts/µL. Hydroxyurea for blast count control is permitted before starting treatment and up to maximum of 10 days after starting treatment on the study. The WBC need not reach 50,000/µL to start hydroxyurea during protocol; the decision to start hydroxyurea during this time is at the discretion of the treating physician
* Active, uncontrolled infection; subjects with infection under active treatment and controlled with antimicrobials are eligible
* Pregnant women
* Uncontrolled undercurrent illness including, but not limited to, symptomatic congestive heart failure, unstable angina pectoris, uncontrolled active seizure disorder, or psychiatric illness/social situations that per site Principal Investigator's judgment would limit compliance with study requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2021-06-11 (Actual); Primary Completion 2025-05-22 (Actual); Study Completion 2025-05-22 (Actual)

PRIMARY OUTCOMES:
Cohort A response rate | through study completion, an average of 1 year
  The rate of achievement of CR+CRh after the first 2 cycles of blinatumomab in Cohort A subjects
Cohort B response rate | through study completion, an average of 1 year
  The rate of achievement of MRD-negativity (< 0.01%) after the first 2 cycles of blinatumomab in Cohort B subjects

SECONDARY OUTCOMES:
Cohort A survival | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months
  To evaluate the following outcomes in subjects with R/R CD19-positive MPAL
  * Achievement of MRD < 0.01% within 2 cycles of treatment with blinatumomab
  * Relapsed free survival (RFS)
  * Event free survival (EFS)
  * Overall survival (OS)
  * Proceeding to allogeneic hematopoietic stem cell transplantation (allo-HSCT) after blinatumomab treatment
  * Overall incidence and severity of adverse events (AEs)
  * CD19-negative and CD19-positive relapse post-blinatumomab
  * The type of lineage switch, as applicable, post-blinatumomab
  * CD19 expression in CSF relapse following blinatumomab, as applicable
  * CAR T-cell treatment of subjects with CSF relapse following blinatumomab and those subjects' outcomes, as applicable
Cohort B survival | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months
  To evaluate the following outcomes in subjects with CD19-positive MPAL in CR/CRh/CRi/CRp after at least one chemotherapy block of standard ALL or AML treatment and detectable MRD at a level of ≥ 0.1% using an assay with a minimum sensitivity of 0.01%
  * Achievement of undetectable MRD (< 0.01%) within one cycle of blinatumomab treatment
  * RFS
  * OS
  * Proceeding to allo-HSCT after blinatumomab treatment
  * Overall incidence and severity of AEs

OTHER OUTCOMES:
CD 19 measurement | through study completion, an average of 1 year
  - Measurement of CD19 trafficking, as a potential mechanism of resistance to blinatumomab by performing flow cytometry, immunohistochemical staining, next generation mRNA sequencing of CD19, CD81, and CD21 exons
CD3-positive measurement | through study completion, an average of 1 year
  - Measurement of CD3-positive T-cells subset as well as function/activity to assess T-cell exhaustion
Leukemic blasts evaluation | through study completion, an average of 1 year
  - Evaluate changes to immunophenotypic characteristics of leukemic blasts in subjects whose disease do not respond to blinatumomab
Subject response evaluation | through study completion, an average of 1 year
  - Evaluate subject responses according to disease-specific features in blasts such as chromosomal amplifications and rearrangements as well as somatic mutations as necessary

CONTACTS AND LOCATIONS:
Overall Officials: Vu Duong, MD, Principal Investigator — University of Maryland, Baltimore
Locations (1):
- Greenebaum Cancer Center at University of Maryland Medical Center, Baltimore, Maryland, United States